CLINICAL TRIAL: NCT04379843
Title: The Efficacy of Implementing a Treatment Algorithm in Managing Patent Ductus Arteriosus (PDA) in the Extremely Low Birth Weight Neonatal Population.
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Collaborators: Banner University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 591107730; 591198726 (Other: MEDNAX CREQS)
Record Dates: First submitted 2020-04-24; First posted 2020-05-08 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: PDA; Low; Birthweight, Extremely (999 Grams or Less)
MeSH Terms: conditions — Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate whether utilizing a standardized patent ductus arteriosus (PDA) treatment algorithm in managing ELBW (extremely low birth weight) neonates ≤1000 grams (g) improves clinical outcomes and helps prevent undesirable side effects from PDAs.

DETAILED DESCRIPTION:
The treatment of PDAs (patent ductus arteriosus) in both the premature and term neonatal population has been the source of thorough research for decades. Common treatment pathways include supportive care, pharmaceutical treatment (via indomethacin, ibuprofen, or acetaminophen), and surgical correction. Many PDAs self-resolve, some are not detected to adulthood, and others may never be discovered. However, determining which neonates with PDAs require pharmaceutical versus surgical management, and which can be managed with supportive care, can be difficult to differentiate. A standardized neonatal PDA treatment algorithm, one that assesses clinical significance, echocardiogram findings, and systemic PDA effects, and one that recommends the optimal treatment course based on these findings, would be helpful in medical management of neonatal PDAs in the ELBW (extremely low birth weight) population.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the BUMCP and CCMC NICUs with a birth weight ≤1000g and an echocardiogram-confirmed PDA, regardless of GA.

Exclusion Criteria:

* Patients who have serious comorbidities that are not directly related to their symptomatic PDA will be excluded (chromosomal abnormalities, serious kidney pathology, other hemodynamically significant heart defects, or serious comorbidities at the researcher's discretion). This will allow the researchers to better determine the efficacy of the treatment algorithm, without the results being confounded by unusual comorbidities.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 100-125 infants ≤1000g with a PDA are born or admitted each year between the BUMCP and CCMC NICUs. Including ELBW neonates over a space of four years will yield a sample size of up to 500, which should be large enough determine how effective the PDA algorithm has been.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
To determine whether using a standardized PDA treatment algorithm improves clinical outcomes in the ELBW population (≤1000 g) with a documented PDA. | 30 days
  - Number of ventilation days {requirement of respiratory support of nasal continuous positive airway pressure (CPAP) or greater}

SECONDARY OUTCOMES:
To determine whether using a standardized treatment algorithm helps prevent undesirable side effects from symptomatic PDAs. | 30 days
  Average length of hospital stay
To determine whether using a standardized treatment algorithm helps prevent undesirable side effects from symptomatic PDAs. | 30 days
  Average weight gain (g/day from birth to discharge)
To determine whether using a standardized treatment algorithm helps prevent undesirable side effects from symptomatic PDAs. | 30 days
  Incidence of bronchopulmonary dysplasia (BPD)
To determine whether using a standardized treatment algorithm helps prevent undesirable side effects from symptomatic PDAs. | 30 days
  Incidence of pulmonary effusion/hemorrhage
To determine whether using a standardized treatment algorithm helps prevent undesirable side effects from symptomatic PDAs. | 30 days
  Incidence of NEC
To determine whether using a standardized treatment algorithm helps prevent undesirable side effects from symptomatic PDAs. | 30 days
  Need for home oxygen (O2) (excluding for high altitude needs at home)
To determine whether using a standardized treatment algorithm helps prevent undesirable side effects from symptomatic PDAs. | 30 days
  Mortality rate
To determine whether using a standardized treatment algorithm helps prevent undesirable side effects from symptomatic PDAs. | 30 days
  Incidence of PDA ligation

OTHER OUTCOMES:
For the group of subjects born after the implementation of the PDA algorithm, a determination will be made as to if the algorithm was followed appropriately. | 30 days
  Review of the subject's chart to determine if treatment algorithm was followed appropriately.
For the group of subjects born after the implementation of the PDA algorithm, a determination will be made as to if the algorithm was followed appropriately. | 30 days
  Calculate compliance rate of algorithm among patients with PDAs.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Banner Cardon Children's Medical Center, Mesa, Arizona
  - Banner - University Medical Center Phoenix, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No